CLINICAL TRIAL: NCT02924857
Title: A Randomized Trial to Confirm the Safety and Effectiveness of Chocolate Touch™ Paclitaxel Coated Balloon Catheter, in Above the Knee Lesions
Brief Title: The Chocolate Touch Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TriReme Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLP788
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Artery Disease (PAD); Ischemia; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Ischemia; Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Test Group (Chocolate Touch) (Experimental): * The diameter of the Chocolate Touch should correspond to the diameter of the vessel for treatment with a balloon to artery ratio of 1.1:1.
  * The Chocolate Touch must be inflated to at least nominal pressure. Maintain balloon inflation for a minimum of 2 minutes. The balloon may be inflated as long as required to achieve optimal angioplasty outcome.
  * If delivery is attempted and failed, a new Chocolate Touch should be used for subsequent attempts after pre-dilatation.
  Interventions: Device: Chocolate Touch
- Control Group (Lutonix Drug Coated Balloon) (Active Comparator): * Never inflate the Lutonix® Drug Coated Balloon (DCB)prior to reaching the target lesion.
  * The Lutonix® Catheter should be advanced to the target site as fast as possible (i.e. 30 seconds) and immediately inflated to appropriate pressure to ensure full wall apposition (balloon to artery ratio of >1:1).
  * If the deployment of the Lutonix® Catheter exceeds 3 minutes, the catheter requires placement with a new unit.
  * Maintain balloon inflation for a minimum of 2 minutes (120 seconds). The balloon may be inflated as long as required by standard of care to achieve a good angioplasty outcome.
  Interventions: Device: Lutonix Drug Coated Balloon

INTERVENTIONS:
Device: Chocolate Touch — The Chocolate Touch™ Paclitaxel Coated Balloon Catheter is indicated for balloon dilatation, after appropriate vessel preparation as needed, of lesions in native superficial femoral or popliteal arteries up to 18 cm in length that are appropriate for angioplasty with balloon diameters from 3.5 mm to 6.0mm.
  Other Names: Chocolate Touch™ Paclitaxel Coated Balloon Catheter
  Arms: Test Group (Chocolate Touch)
Device: Lutonix Drug Coated Balloon — The Lutonix® 035 Drug Coated Balloon Catheter is indicated for improving luminal diameter for the treatment of obstructive de novo or non-stented restenotic lesions (≤ 18 cm in length) in native femoropopliteal arteries having reference vessel diameters of 4 mm to 6 mm.
  Other Names: LUTONIX® 035 Drug Coated Balloon Catheter
  Arms: Control Group (Lutonix Drug Coated Balloon)

SUMMARY:
The Chocolate Touch study is a randomized, multi-center, prospective, adaptive study, designed to show sufficient safety and effectiveness of the Chocolate Touch™ for use in superficial femoral or popliteal arteries with the intention of obtaining regulatory approval to market this device in the United States

DETAILED DESCRIPTION:
The primary objective of the Chocolate Touch study is to demonstrate non-inferior safety and non-inferior effectiveness of the Chocolate Touch™ compared to the Lutonix® drug coated balloon catheter. These data are intended to show safety and effectiveness of the Chocolate Touch sufficient to support regulatory approval to market this device in the United States for use in superficial femoral or popliteal arteries.

Study success is defined as statistical demonstration of the non-inferiority hypothesis tests for both the primary safety and effectiveness hypothesis.

PMA P210039 approval has been granted on 11/04/2022. The study is now in the post-approval phase.

ELIGIBILITY:
Inclusion Criteria

General:

1. Minimum of 18 years of age
2. Intermittent claudication or ischemic rest pain (Rutherford 2-4)
3. Life Expectancy >2 years
4. Patient has agreed to follow-up requirements and given informed consent

   Angiographic:
5. Lesion successfully crossed with a guidewire
6. Lesion in the SFA or popliteal artery defined as a lesion with a proximal origin >10 mm from SFA origin (deep femoral artery) and a distal end above the knee joint (at least 3 cm above bottom of the femur - P1).
7. Target Lesion ≥70% stenosis in the SFA or popliteal arteries
8. Reference Vessel Diameter (RVD) between 4.0 & 6.0mm and within treatment range of Chocolate Touch to be used 1.1:1 at the Target Lesion
9. Target Lesion ≤180mm that consists of no more than two adjacent lesions (≤ 25mm apart) and is able to be completely covered with inflation of no more than two assigned balloons (with minimum of >5mm overlap to the area covered by the first balloon). (Note: Adjacent or tandem target lesions must be treated as a single lesion.)
10. Angiographic evidence of distal run-off demonstrated by at least one patent tibial vessel without evidence of significant (≥70%) stenosis from origin to ankle
11. In-flow vessel without significant stenosis (≥70%) or successful treatment (≤30% residual stenosis with no complications) of a diseased vessel. Note: treatment of contralateral iliac is permissible.

Exclusion Criteria

General:

1. Acute limb ischemia, or patient indicated for thrombolytic therapy
2. Planned surgical or interventional procedures within 30 days after study procedure.
3. Non-target lesion concurrent interventions involving a re-entry device, atherectomy, laser, or ablation procedures, the use of a drug eluting stent, or, treatment with any other drug coated balloon.
4. Myocardial infarction or stroke within 30 days prior to the procedure
5. Known intolerance to required medications, contrast media that cannot be adequately premedicated, nitinol, or Paclitaxel
6. Known impaired Renal Function that could have an impact on contrast tolerance with GFR ≤ 30 ml/min per 1.73 m2 and/or elevated serum creatinine >2.5mg/dL (220µmol/L) or on dialysis.
7. Known bleeding disorder, or on dialysis, or uncontrolled hypercoagulable disorder
8. Non-atherosclerotic lesion (e.g. vasculitis or Berger's disease)
9. Female who is pregnant or intends to be pregnant during study
10. Patient is enrolled in another investigational clinical study or was previously enrolled in this study

    Angiographic:
11. Presence of perforation, dissection (Type D or worse) or other injury in target vessel at time of enrollment
12. Severe Calcification at the target lesion (defined as angiographic evidence of dense calcification present on both sides of the vessel wall on two orthogonal views and that extends >50 continuous mm in length).
13. Previous bypass graft, stent at target vessel (must be greater than 20mm from target lesion), or iliac stent that cannot permit crossing by the treatment balloon within the introducer sheath (Note: In-stent restenosis is not allowed.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
True Drug Coated Balloon Success | 12 months
  A composite endpoint that requires patients to achieve Primary Patency (Peak systolic velocity ratio <2.4 without the need for clinically driven target lesion revascularization) in the absence of a clinically driven bail-out stent (core lab adjudicated).
Freedom from Major Adverse Events | 12 months
  Composite of target-limb-related death, major amputation of the target limb, and clinically driven re-intervention of the target limb.

SECONDARY OUTCOMES:
By Angiographic Core Lab Review (Acute) | 1 hour
  Procedural Success: Defined as the success of the therapy to achieve <30% diameter stenosis without a flow-limiting dissection or the need for a stent
By Duplex Ultrasound Core Lab Review | 6, 12, 24, & 36 months
  Patency
By Clinical Assessment | 6, 12, 24, & 36 months
  Occurrence of relevant Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Shishehbor, DO, Principal Investigator — Cleveland Medical Center, Cleveland, Ohio; Thomas Zeller, MD, Principal Investigator — Universitat Herzzentrum, Bad Krozingen, Germany
Locations (20):
- United States (15):
  - Cardiac and Vascular Institute, Gainesville, Florida
  - Mt. Sinai - Miami, Miami Beach, Florida
  - Emory University, Atlanta, Georgia
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Michigan Outpaitient Vascular Institution, Dearborn, Michigan
  - Jackson Heart, Jackson, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Mt. Sinai Heart, New York, New York
  - Columbia University Medical Center / NewYork Presbyterian Hospital, New York, New York
  - Univeristy Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Penn State Health Holy Spirit Medical Center, Camp Hill, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - MIssion Research, New Braunfels, Texas
  - Swedish Medical Center, Seattle, Washington
- Austria (2):
  - Medical University of Graz - LKH Univ.-Klinikum Graz, Graz
  - Angiologie - Hansuchkrankenhaus, Vienna
- Universitat Herz-Zentrum, Bad Krozingen, Germany
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Selvin E, Erlinger TP. Prevalence of and risk factors for peripheral arterial disease in the United States: results from the National Health and Nutrition Examination Survey, 1999-2000. Circulation. 2004 Aug 10;110(6):738-43. doi: 10.1161/01.CIR.0000137913.26087.F0. Epub 2004 Jul 19. PMID 15262830
- [Background] Hirsch AT, Criqui MH, Treat-Jacobson D, Regensteiner JG, Creager MA, Olin JW, Krook SH, Hunninghake DB, Comerota AJ, Walsh ME, McDermott MM, Hiatt WR. Peripheral arterial disease detection, awareness, and treatment in primary care. JAMA. 2001 Sep 19;286(11):1317-24. doi: 10.1001/jama.286.11.1317. PMID 11560536
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892
- [Background] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447
- [Background] Scheinert D, Duda S, Zeller T, Krankenberg H, Ricke J, Bosiers M, Tepe G, Naisbitt S, Rosenfield K. The LEVANT I (Lutonix paclitaxel-coated balloon for the prevention of femoropopliteal restenosis) trial for femoropopliteal revascularization: first-in-human randomized trial of low-dose drug-coated balloon versus uncoated balloon angioplasty. JACC Cardiovasc Interv. 2014 Jan;7(1):10-9. doi: 10.1016/j.jcin.2013.05.022. PMID 24456716
- [Background] Schmidt A, Piorkowski M, Werner M, Ulrich M, Bausback Y, Braunlich S, Ick H, Schuster J, Botsios S, Kruse HJ, Varcoe RL, Scheinert D. First experience with drug-eluting balloons in infrapopliteal arteries: restenosis rate and clinical outcome. J Am Coll Cardiol. 2011 Sep 6;58(11):1105-9. doi: 10.1016/j.jacc.2011.05.034. PMID 21884945
- [Background] Werk M, Albrecht T, Meyer DR, Ahmed MN, Behne A, Dietz U, Eschenbach G, Hartmann H, Lange C, Schnorr B, Stiepani H, Zoccai GB, Hanninen EL. Paclitaxel-coated balloons reduce restenosis after femoro-popliteal angioplasty: evidence from the randomized PACIFIER trial. Circ Cardiovasc Interv. 2012 Dec;5(6):831-40. doi: 10.1161/CIRCINTERVENTIONS.112.971630. Epub 2012 Nov 27. PMID 23192918
- [Background] Schnorr B, Kelsch B, Cremers B, Clever YP, Speck U, Scheller B. Paclitaxel-coated balloons - Survey of preclinical data. Minerva Cardioangiol. 2010 Oct;58(5):567-82. PMID 20948503
- [Background] Schnorr B, Speck U, Scheller B. Review of clinical data with Paccocath- coated balloon catheters. Minerva Cardioangiol. 2011 Oct;59(5):431-45. PMID 21983304
- [Background] Zeller T, Schmitmeier S, Tepe G, Rastan A. Drug-coated balloons in the lower limb. J Cardiovasc Surg (Torino). 2011 Apr;52(2):235-43. PMID 21460774
- [Background] Morikawa T, Yoshida M. A useful testing strategy in phase III trials: combined test of superiority and test of equivalence. J Biopharm Stat. 1995 Nov;5(3):297-306. doi: 10.1080/10543409508835115. PMID 8580930
- [Background] Shishehbor MH, Zeller T, Werner M, Brodmann M, Parise H, Holden A, Lichtenberg M, Parikh SA, Kashyap VS, Pietras C, Tirziu D, Ardakani S, Beschorner U, Krishnan P, Niazi KA, Wali AU, Lansky AJ. Randomized Trial of Chocolate Touch Compared With Lutonix Drug-Coated Balloon in Femoropopliteal Lesions (Chocolate Touch Study). Circulation. 2022 May 31;145(22):1645-1654. doi: 10.1161/CIRCULATIONAHA.122.059646. Epub 2022 Apr 4. PMID 35377157
- [Background] Bohme T, Zeller T, Shishehbor MH, Werner M, Brodmann M, Parise H, Holden A, Lichtenberg M, Parikh SA, Kashyap VS, Pietras C, Tirziu D, Beschorner U, Krishnan P, Niazi KA, Wali AU, Lansky AJ. Chocolate Touch Versus Lutonix Drug-Coated Balloon for Femoropopliteal Lesions in Diabetes: The Chocolate Touch Study. J Endovasc Ther. 2025 Apr;32(2):414-422. doi: 10.1177/15266028231179589. Epub 2023 Jun 14. PMID 37314243